CLINICAL TRIAL: NCT02684448
Title: A Retrospective Multi-Center Study for Evaluation of Clinical Outcomes in Inguinal Hernia Repair
Brief Title: Evaluation of Clinical Outcomes in Robotic-Assisted Inguinal Hernia Repair
Status: Completed | Type: Observational
Sponsor: Intuitive Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: ISI-IHR-2015-001
Record Dates: First submitted 2016-02-12; First posted 2016-02-18 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Hernia, Inguinal; Hernia, Inguinal, Direct; Hernia, Inguinal, Indirect
MeSH Terms: conditions — Hernia, Inguinal | interventions — Herniorrhaphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Robotic-Assisted Inguinal Hernia Repair: Subjects who have undergone robotic-assisted (da Vinci) inguinal hernia repair from the initiation of robotic-assisted hernia repair at site through December 2015.
  Interventions: Procedure: Inguinal Hernia Repair
- Open Inguinal Hernia Repair: Subjects who have undergone open inguinal hernia repair from the day prior to initiation of robotic-assisted hernia repair through 5 years prior to initiation.
  Interventions: Procedure: Inguinal Hernia Repair

INTERVENTIONS:
Procedure: Inguinal Hernia Repair — Inguinal (unilateral or bilateral) hernia repair
  Other Names: Herniorrhaphy

SUMMARY:
This multi-center, retrospective data collection study will evaluate the feasibility, safety and performance of the da Vinci® surgical system for patients who have undergone robotic-assisted inguinal hernia repair, as well as provide information about the learning curve associated with robotic-assisted (da Vinci®) inguinal hernia repair.

In addition, this retrospective data collection study will evaluate the perioperative outcomes of robotic-assisted (da Vinci®) inguinal hernia repair and compare perioperative outcomes with those associated with open hernia repair by the same participating surgeon.

DETAILED DESCRIPTION:
This study is a retrospective data collection from existing medical records, is observational in nature and is designed to evaluate feasibility, safety and performance of the da Vinci® surgical system for patients who have undergone inguinal hernia repair surgery during the time period from initiation of robotic-assisted surgery to 30 days prior to study initiation (IRB approval and fully executed data collection agreement) for approximately 500 subjects. Any inguinal hernia repair procedure that uses the da Vinci® surgical system at any point will be collected.

This data will be compared with data associated with open inguinal hernia repairs performed by the same surgeons from a period of 5 years prior to the initiation of robotic surgery at each participating institution until 30 days prior to study initiation. Sites will collect data from consecutive open inguinal hernia repair cases starting with the day prior to the 1st robotic-assisted inguinal hernia repair, and continue collecting data until the number of open inguinal hernia repair cases is equivalent to the number of robotic-assisted inguinal hernia repair cases, or until the open repair procedure date reaches 5 years prior to the 1st robotic-assisted inguinal hernia repair case.

Data collected will include, but is not limited to, the following:

1. Demographics and baseline/pre-operative clinical parameters: Gender, age, BMI, comorbidities, smoking history, prior hernia history, prior abdominal surgery history, hernia description
2. Intraoperative parameters: procedure details related to repair, operative time, conversions to open, blood loss, intraoperative complications
3. Post-operative through discharge : length of hospital stay, post-operative complications
4. Post-operative information regarding complications, readmissions and reoperations through 30 days post-discharge.
5. Hernia Recurrence, if available

The total duration for this study will be approximately 12 months

ELIGIBILITY:
Inclusion Criteria:

all patients who have undergone inguinal hernia repair using either an open technique or a robotic-assisted (da Vinci®) approach

Eligible subjects must have had their inguinal hernia repair completed according to the following timeframes for inclusion:

1. Robotic-assisted (da Vinci®) hernia repair - all consecutive robotic cases from the initiation of robotic -assisted inguinal hernia repair at each institution until 30 days prior to the date of study initiation (IRB approval and fully executed contract).
2. Open hernia repair - all consecutive open hernia repair cases from the day prior to the 1st da Vinci® inguinal hernia repair until the number of open repair cases collected is equivalent to the number of da Vinci® cases entered, or the date 5 years pre-robotic initiation is reached.

Exclusion Criteria:

* Subjects who have undergone robotic-assisted or open inguinal hernia repair outside of required timeframe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who have undergone robotic-assisted inguinal hernia repair or open hernia repair per specified time frame described in inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 1258 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Number of complications observed intraoperatively through 30-days | Intraoperative through 30-days follow-up

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Progressive Surgical Associates/Silver Cross Hospital, New Lenox, Illinois
  - Rochester General Hospital, Rochester, New York

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Derived] Dickens EO, Kolachalam R, Gonzalez A, Richardson C, D'Amico L, Rabaza J, Gamagami R. Does robotic-assisted transabdominal preperitoneal (R-TAPP) hernia repair facilitate contralateral investigation and repair without compromising patient morbidity? J Robot Surg. 2018 Dec;12(4):713-718. doi: 10.1007/s11701-018-0815-4. Epub 2018 Apr 30. PMID 29713930